CLINICAL TRIAL: NCT07357259
Title: Delayed Pelvic Imaging With [68]Ga-PSMA PET/CT in a Patient With High-risk Prostate Cancer.
Acronym: SPIR202302
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Michela Moscarino, Principal Investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SPIR202302
Record Dates: First submitted 2025-12-04; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: High-risk Prostate Cancer
Keywords: PET/CT; [68]Ga - PSMA; Delay CT scan; Radiation Dose Optimization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (A) (No Intervention): Participants will undergo the conventional [⁶⁸Ga]Ga-PSMA PET/CT protocol, which includes a standard whole-body PET/CT performed 60 minutes post-injection and a delayed pelvic PET/CT as per current clinical practice (PET + CT).
- Intervention Group (B) (Experimental): Participants will undergo:
  * Standard whole-body PET/CT at 60 minutes, followed by
  * A delayed pelvic PET-only acquisition at 90 minutes, reconstructed using the CT obtained during the initial whole-body acquisition.
  Interventions: Diagnostic Test: Intervention Group

INTERVENTIONS:
Diagnostic Test: Intervention Group — Matching of delayed PET images with the standard CT scan
  Arms: Intervention Group (B)

SUMMARY:
Recent evidence suggests that both standard-time and delayed-time [⁶⁸Ga]Ga-PSMA PET acquisitions can reveal clinically relevant findings, and neither phase should be excluded a priori in routine practice. This study evaluates a streamlined dual-phase protocol consisting of:

* A standard whole-body PET/CT acquisition performed 60 minutes after radiotracer administration.
* A delayed pelvic PET-only acquisition performed 90 minutes post-injection, reconstructed using the attenuation-correction CT (CT/AC) obtained from the initial whole-body scan.

Because the prostate gland and pelvic lymph nodes exhibit minimal physiological mobility, accurate PET-CT anatomical correspondence can be maintained through careful patient repositioning, without repeating the CT scan.

The main advantage of this protocol is a reduction in patient radiation exposure, as the delayed phase does not require a second CT scan. It also reduces in-department time and maintains diagnostic quality of PET interpretation, provided that the PET-CT alignment remains acceptable.

This method may additionally enhance workflow efficiency in the Nuclear Medicine Unit by allowing early identification-based on predefined clinical parameters-of patients most likely to benefit from delayed pelvic imaging.

DETAILED DESCRIPTION:
This study evaluates a modified dual-phase [⁶⁸Ga]Ga-PSMA PET/CT protocol designed to reduce radiation exposure and streamline workflow while maintaining diagnostic quality in the assessment of prostate cancer. Conventional imaging often includes a standard whole-body PET/CT acquisition at approximately 60 minutes post-injection followed by a delayed pelvic PET/CT, which can provide additional lesion detectability but requires a second CT scan. The additional CT increases both radiation dose and examination duration.

The proposed protocol replaces the delayed CT with a PET-only pelvic acquisition performed 90 minutes post-injection. Delayed PET images are reconstructed and attenuation-corrected using the CT dataset obtained during the initial whole-body acquisition. This approach is feasible because pelvic structures relevant to prostate cancer-such as the prostate gland and pelvic lymph nodes-exhibit limited physiological motion compared with intraperitoneal organs, allowing reliable PET-CT anatomical correspondence through optimized patient repositioning.

The study adopts a randomized, two-arm design including patients undergoing staging for newly diagnosed prostate cancer or evaluation of biochemical recurrence. Randomization is stratified by prior radical prostatectomy to account for potential anatomical variability. The control arm follows the standard clinical workflow with both standard and delayed PET/CT acquisitions. The intervention arm undergoes standard whole-body PET/CT at 60 minutes and delayed PET-only imaging at 90 minutes.

Anatomical matching between delayed PET images and the CT dataset will be independently evaluated by three Medical Imaging Technologists (TSRM1, TSRM2, TSRM3) across three blinded reading sessions. Each rater will score image alignment using a standardized 1-5 Likert scale. The primary endpoint is the quality of PET-CT matching, assessed through Fleiss' kappa statistics to quantify interrater agreement and compare matching performance between the two imaging workflows.

Secondary objectives examine the potential reduction in radiation exposure, measured through CTDIvol and DLP values obtained from the CT Dose Report, and the impact on patient experience and departmental efficiency. Patient-perceived waiting time and comfort will be assessed through a short questionnaire administered after the examination, while objective in-department duration will be extracted from institutional scheduling records.

If effective, the streamlined protocol may support broader adoption of CT-free delayed pelvic imaging by demonstrating that optimized technologist-led positioning can maintain diagnostic interpretability while improving patient-centered outcomes and reducing overall radiation burden.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed prostate cancer undergoing staging, or
* Biochemical recurrence following prior radical-intent therapy (surgery and/or radiotherapy), or
* High-risk prostate cancer, defined as Gleason Score ≥ 8 or PSA ≥ 20 ng/mL.
* Written informed consent and authorization for personal data processing.

Exclusion Criteria:

* Genitourinary comorbidities that could interfere with imaging or interpretation.
* Intermediate- or low-risk prostate cancer.
* Delayed acquisition performed on a PET/CT scanner different from the standard acquisition.
* Additional PET/CT required due to artifacts compromising diagnostic quality (e.g., urinary retention, excessive motion).
* Patients previously enrolled who require repeat PET/CT as a new visit.
* Inability to provide informed consent or impaired decision-making capacity.
* Known hypersensitivity to the radiopharmaceutical or its components.
* Contraindications to PET/CT (e.g., severe claustrophobia, morbid obesity, inability to cooperate).

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Matching Quality of Delayed PET with Standard CT | Up to completion of the study, on average 1 year.
  Evaluation of the actual matching accuracy between delayed PET images-reconstructed and attenuation-corrected using the dedicated CT/AC dataset-and the standard CT scan within the new procedural approach to [68]Ga-PSMA PET/CT. Three Technologist of Medical Imaging (TSRM1, TSRM2, TSRM3) will evaluate the images independently, in a blinded manner, at three separate time points (t1, t2, t3).
  The registration accuracy between delayed PET images and the standard CT scan will be evaluated using a qualitative questionnaire based on the evaluators' professional experience (minimum of five years in Nuclear Medicine). Image registration will be scored on a 5-point ordinal scale, ranging from 1 (complete mismatch) to 5 (perfect registration).
  Unit of Measure: 5-point ordinal scale (1-5)

SECONDARY OUTCOMES:
Radiation Dose Optimization | Up to completion of study, on average 1 year.
  Change in CTDIvol (Computed Tomography Dose Index volume) in the experimental arm. CTDIvol (mGy) will be used to assess changes in radiation dose related to the experimental protocol.
  Unit of Measure:
  Milligray (mGy)
Patient Throughput and Experience | Up to completion of study, on average 1 year.
  Comparison of patient experience in the Nuclear Medicine Unit between the two study groups. Patient experience will be evaluated using a structured, patient-reported questionnaire at the end of the [68]Ga-PSMA PET/CT examination, based on the perceived quality of staff information regarding waiting times.
  Unit of Measure:
  - Patient experience: 5-level ordinal scale (Very poor → Excellent)

OTHER OUTCOMES:
Radiation Dose Optimization | Up to completion of the study, on average 1 year.
  Change in Dose Length Product (DLP) in the experimental arm. DLP (mGy * cm) will be used to assess changes in cumulative radiation dose along the scan length associated with the experimental protocol.
  Unit of Measure:
  Milligray·centimeter (mGy·cm)
  Notes:
  This measure is part of Secondary Outcome 2: Radiation Dose Optimization
Radiation Dose Optimization | Up to completion of the study, on average 1 year.
  Change in Effective Dose in the experimental arm. Effective dose (mSv) will be estimated to evaluate overall patient radiation exposure associated with the experimental protocol.
  Unit of Measure:
  Millisievert (mSv)
  Notes:
  This measure is part of Secondary Outcome 2: Radiation Dose Optimization
Patient Throughput and Experience | Up to completion of the study, on average 1 year
  Comparison of perceived waiting time in the Nuclear Medicine Unit between the two study groups. Perceived waiting time will be reported by patients for each questionnaire item in minutes (m).
  Minutes (categorical ranges per questionnaire item, e.g., <5, 5-10, 10-15, >15)
  Notes: This parameter is part of the single secondary outcome 3: 3. Patient Throughput and Experience

CONTACTS AND LOCATIONS:
Overall Officials: Michela Moscarino, Technician, Principal Investigator — IRCCS Università di Bologna, Policlinico di Sant'Orsola
Locations (1):
- IRCCS - Policlinico Universitario di Sant'Orsola, Bologna, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoffmann MA, Buchholz HG, Wieler HJ, Rosar F, Miederer M, Fischer N, Schreckenberger M. Dual-Time Point [68Ga]Ga-PSMA-11 PET/CT Hybrid Imaging for Staging and Restaging of Prostate Cancer. Cancers (Basel). 2020 Sep 28;12(10):2788. doi: 10.3390/cancers12102788. PMID 32998432
- [Background] Rahbar K, Afshar-Oromieh A, Bogemann M, Wagner S, Schafers M, Stegger L, Weckesser M. 18F-PSMA-1007 PET/CT at 60 and 120 minutes in patients with prostate cancer: biodistribution, tumour detection and activity kinetics. Eur J Nucl Med Mol Imaging. 2018 Jul;45(8):1329-1334. doi: 10.1007/s00259-018-3989-0. Epub 2018 Mar 14. PMID 29541812
- [Background] Haupt F, Dijkstra L, Alberts I, Sachpekidis C, Fech V, Boxler S, Gross T, Holland-Letz T, Zacho HD, Haberkorn U, Rahbar K, Rominger A, Afshar-Oromieh A. 68Ga-PSMA-11 PET/CT in patients with recurrent prostate cancer-a modified protocol compared with the common protocol. Eur J Nucl Med Mol Imaging. 2020 Mar;47(3):624-631. doi: 10.1007/s00259-019-04548-5. Epub 2019 Nov 1. PMID 31673789
- [Background] Derlin T, Weiberg D, von Klot C, Wester HJ, Henkenberens C, Ross TL, Christiansen H, Merseburger AS, Bengel FM. 68Ga-PSMA I&T PET/CT for assessment of prostate cancer: evaluation of image quality after forced diuresis and delayed imaging. Eur Radiol. 2016 Dec;26(12):4345-4353. doi: 10.1007/s00330-016-4308-4. Epub 2016 Mar 24. PMID 27011373
- [Background] Beheshti M, Manafi-Farid R, Geinitz H, Vali R, Loidl W, Mottaghy FM, Langsteger W. Multiphasic 68Ga-PSMA PET/CT in the Detection of Early Recurrence in Prostate Cancer Patients with a PSA Level of Less Than 1 ng/mL: A Prospective Study of 135 Patients. J Nucl Med. 2020 Oct;61(10):1484-1490. doi: 10.2967/jnumed.119.238071. Epub 2020 Feb 14. PMID 32060214
- [Background] Fonti R, Conson M, Del Vecchio S. PET/CT in radiation oncology. Semin Oncol. 2019 Jun;46(3):202-209. doi: 10.1053/j.seminoncol.2019.07.001. Epub 2019 Jul 26. PMID 31378377
- [Background] Fanti S, Minozzi S, Antoch G, Banks I, Briganti A, Carrio I, Chiti A, Clarke N, Eiber M, De Bono J, Fizazi K, Gillessen S, Gledhill S, Haberkorn U, Herrmann K, Hicks RJ, Lecouvet F, Montironi R, Ost P, O'Sullivan JM, Padhani AR, Schalken JA, Scher HI, Tombal B, van Moorselaar RJA, Van Poppel H, Vargas HA, Walz J, Weber WA, Wester HJ, Oyen WJG. Consensus on molecular imaging and theranostics in prostate cancer. Lancet Oncol. 2018 Dec;19(12):e696-e708. doi: 10.1016/S1470-2045(18)30604-1. PMID 30507436
- [Background] Purohit RS, Shinohara K, Meng MV, Carroll PR. Imaging clinically localized prostate cancer. Urol Clin North Am. 2003 May;30(2):279-93. doi: 10.1016/s0094-0143(02)00184-2. PMID 12735504
- [Background] Schroder FH, Hugosson J, Roobol MJ, Tammela TL, Ciatto S, Nelen V, Kwiatkowski M, Lujan M, Lilja H, Zappa M, Denis LJ, Recker F, Berenguer A, Maattanen L, Bangma CH, Aus G, Villers A, Rebillard X, van der Kwast T, Blijenberg BG, Moss SM, de Koning HJ, Auvinen A; ERSPC Investigators. Screening and prostate-cancer mortality in a randomized European study. N Engl J Med. 2009 Mar 26;360(13):1320-8. doi: 10.1056/NEJMoa0810084. Epub 2009 Mar 18. PMID 19297566